CLINICAL TRIAL: NCT04607486
Title: Reliability Study of a 3D Free-hand Ultrasonography Technique (3DfUS) in Combination With Instrumented Spasticity Assessment (ISA) for the Lower Limb in Chronic First-ever Stroke Patients.
Brief Title: Investigation of Changes in Lower Limb Muscles After Cerebrovascular Accident
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S60153
Record Dates: First submitted 2020-08-06; First posted 2020-10-29 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CVA and spasticity: Adults with first-ever chronic CVA and leg spasticity
  Interventions: Diagnostic Test: 3DfUS and IPSA of leg muscles
- CVA without spasticity: Control group
  Interventions: Diagnostic Test: 3DfUS and IPSA of leg muscles
- healthy subjects: Control group
  Interventions: Diagnostic Test: 3DfUS and IPSA of leg muscles

INTERVENTIONS:
Diagnostic Test: 3DfUS and IPSA of leg muscles — 1. 3DfUS technique enhances a conventional 2D US device into a platform capable of reconstructing 3D anatomical data sets.
  2. IPSA for quantification of hyper-resistance and its underlying components. The sensors in the IPSa include gyroscopes and accelerometers to measure joint angle and angular velocity, EMG to measure muscle activity, and a 3 degrees-of freedom force sensor to measure torque applied on the joint.
  3. clinical functional capacity = clinical evaluation of degree of independence, mobility and gait
  Other Names: clinical functional capacity

SUMMARY:
The aim of this study is to investigate lower limb muscles after cerebrovascular accident

DETAILED DESCRIPTION:
The aim of this study is to define and differentiate the changes in MMT properties related to the alterations in muscle tone of the lower limb in first-ever chronic stroke patients by using a 3D free-hand Ultrasonography (3DfUS) technique in combination with an instrumented spasticity assessment (IPSA). In these chronic stroke patients, the spontaneous neurological recovery is stabilized

ELIGIBILITY:
Inclusion Criteria:

* Definition of case population :

  o first ever stroke with spasticity of the lower limb.
* Definition of control :

  * first ever stroke without spasticity of the lower limb
  * healthy aged-matched subjects

Exclusion Criteria:

* Musculoskeletal or neurological problems affecting the lower limb
* Presence of other neurological pathology that could lead to spasticity, ataxia, dystonia
* Cognitive problems that impede measurements
* Severe co-morbidities
* Peripheral spastic medication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with first ever chronic stroke:
  = First ever stroke subjects with established spasticity and without spasticity will be recruited on the stroke rehabilitation unit and outpatient rehabilitation clinic, University Hospital of Leuven.
  Healthy control subjects
  = Healthy age-and gender matched subjects will be recruited among healthy university staff of the University Hospital of Leuven, their family and friends.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Muscle volume | 1 day
  Estimation of muscle volume by 3D freehand ultrasonography.
Muscle and Tendon Length | 1 day
  Estimation of muscle volume by 3D freehand ultrasonography
Echogenicity intensity | 1 day
  Estimation of echogenicity intensity by 3D freehand ultrasonography on an 8-bit greyscale (256 values).
Work [J] derived from the slow stretch | 1 day
  Measurement of Work [J] by Instrumented Spasticity Assessment
Muscle activity EMG [uV] derived from the fast stretch | 1 day
  Measurement of Muscle activity EMG [uV] by Instrumented Spasticity Assessment
Maximal velocity of performance (Vmax [deg/s]) | 1 day
  Measurement of Maximal velocity of performance (Vmax [deg/s]) by Instrumented Spasticity Assessment
Range of motion [deg] for slow stretch | 1 day
  Measurement of Range of motion [deg] by Instrumented Spasticity Assessment
Stiffness [Nm/deg] for slow stretch | 1 day
  Measurement of Stiffness [Nm/deg] by Instrumented Spasticity Assessment
Joint angle of catch [deg] from the fast stretch | 1 day
  Measurement of Joint angle of catch [deg] from the fast stretch by Instrumented Spasticity Assessment
Angle of EMG threshold [deg] from the fast stretch | 1 day
  Measurement of Angle of EMG threshold [deg] by Instrumented Spasticity Assessment
Intensity of catch derived from the fast stretch | 1 day
  Measurement of Intensity of catch by Instrumented Spasticity Assessment

SECONDARY OUTCOMES:
Clinical assessment of spasticity at fast stretch | 1 day
  Estimation of spasticity by Modified Assessment Scale
Clinical assessment of spasticity angle at slow and fast stretch | 1 day
  Estimation of spasticity by Tardieu Scale

OTHER OUTCOMES:
Quantify the impairment caused by a stroke | 1 day
  Evaluation of impairment caused by stroke by National Institute Health Stroke Scale
Assessments of functional independence in daily life in stroke patients and healthy subjects | 1 day
  Evaluation of functional independence in daily life is assessed by the Barthel Index
Assessments of functional status after stroke | 1 day
  Evaluation of functional status after stroke is assessed by the Functional Independence Measure
Assessesment of mobility in stroke patients | 1 day
  Evaluation of mobility after stroke is assessed by the Rivermead Mobility Index
Assessment of transfer skills in stroke patients and healthy subjects | 1 day
  Measurement of functional lower extremity strength and/or identify movement strategies in stroke patients and healthy subjects by The Five Times Sit to Stand Test
Assessment of the motor impairment in lower limbs of stroke patients | 1 day
  Measurement of lower limb strength in stroke patients by the Motricity Index
Assessments of gait speed analysis in stroke patients and healthy subjects. | Measurement of gait speed in stroke patients and healthy subjects by 5-Meter Walk Test at comfortable or self-selected gait speed.
  1 day

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Schillebeeckx, MD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided